CLINICAL TRIAL: NCT06958198
Title: A Phase Ib Age De-escalation, Open Label Study of the Safety and Immunogenicity of the Multi-stage Malaria Vaccine Candidate R21 + RH5.1 + R78C in Matrix-M™ in Adults Aged 18-35 Years and Children Aged 5-17 Months in Burkina Faso
Brief Title: A Study to Assess the Experimental Malaria Vaccines R78C and RH5.1 Combined With R21/Matrix-M (a "Multi-stage" Malaria Vaccine)
Acronym: VAC093
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Wellcome Trust (Other); European Vaccine Initiative (Other); Bundesministerium für Forschung, Technologie und Raumfahrt (BMFTR) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC093
Record Dates: First submitted 2025-04-23; First posted 2025-05-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-04

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — R21 monoclonal antibody; Matrix-M

STUDY DESIGN:
Intervention Model Description: This is a Phase Ib age de-escalation, dose escalation, open label study to assess the safety and immunogenicity of the multi-stage malaria vaccine candidate R21 plus RH5.1 and/or R78C in Matrix-M in adults aged 18-35 years and children aged 5-17 months in Burkina Faso. 8 healthy adults aged 18-35 years and 48 children aged 5-17 months living in a malaria endemic area will be recruited at one site in Burkina Faso. Adults will be recruited into one group receiving the combination of R21 + RH5.1 + R78C in Matrix-M. Children will be recruited into four groups receiving the combination of the three vaccines, R21 + RH5.1/Matrix-M, R21 + R78C/Matrix-M, R21/Matrix-M only or RH5.1 + R78C/Matrix-M only.
  Follow-up will be for 6 months post third vaccination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1(n=8) adults (18-35years) (Experimental): They will receive three doses of 5 µg R21 + 10 µg RH5.1 + 10 µg R78C, administered at Month 0 (Day 0), Month 1 (Day 28), and Month 6 (Day 182), given as an Intramuscular injection to the deltoid region (adults) or anterolateral thigh (children)
  Interventions: Biological: R21; Biological: RH5.1; Biological: R78C; Biological: Matrix-M™
- Group 2 (n=8) Children aged between 5-17months (Experimental): They will receive three doses of 5 µg R21 + 10 µg RH5.1, administered at Month 0 (Day 0), Month 1 (Day 28), and Month 6 (Day 182), given as an Intramuscular injection to the deltoid region (adults) or anterolateral thigh (children)
  Interventions: Biological: R21; Biological: RH5.1; Biological: Matrix-M™
- Group 3 (n=8) children aged between 5-17 months (Experimental): They will receive three doses of 5 µg R21 + 10 µg R78C, administered at Month 0 (Day 0), Month 1 (Day 28), and Month 6 (Day 182), given as an Intramuscular injection to the deltoid region (adults) or anterolateral thigh (children)
  Interventions: Biological: R21; Biological: R78C; Biological: Matrix-M™
- Group 4 (n=8) Children aged between 5-17 months (Experimental): They will receive three doses of 5 µg R21 + 10 µg RH5.1 +10 µg R78C , administered at Month 0 (Day 0), Month 1 (Day 28), and Month 6 (Day 182), given as an Intramuscular injection to the deltoid region (adults) or anterolateral thigh (children)
  Interventions: Biological: R21; Biological: RH5.1; Biological: R78C; Biological: Matrix-M™
- Group 5 (n=8) children aged 5-17 months (Experimental): They will receive three doses of 5 µg R21, administered at Month 0 (Day 0), Month 1 (Day 28), and Month 6 (Day 182), given as an Intramuscular injection to the deltoid region (adults) or anterolateral thigh (children)
  Interventions: Biological: R21; Biological: Matrix-M™
- Group 6 ( n=16) Children 5-17 months (Experimental): They will receive three doses of 10 µg RH5.1 +10 µg R78C, administered at Month 0 (Day 0), Month 1 (Day 28), and Month 6 (Day 182), given as an Intramuscular injection to the deltoid region (adults) or anterolateral thigh (children)
  Interventions: Biological: RH5.1; Biological: R78C; Biological: Matrix-M™

INTERVENTIONS:
Biological: R21 — A protein particle comprising recombinant HBsAg fused to the central repeat and the C-terminus of the circumsporozoite protein
  Arms: Group 1(n=8) adults (18-35years); Group 2 (n=8) Children aged between 5-17months; Group 3 (n=8) children aged between 5-17 months; Group 4 (n=8) Children aged between 5-17 months; Group 5 (n=8) children aged 5-17 months
Biological: RH5.1 — A soluble protein vaccine against the RH5 antigen
  Arms: Group 1(n=8) adults (18-35years); Group 2 (n=8) Children aged between 5-17months; Group 4 (n=8) Children aged between 5-17 months; Group 6 ( n=16) Children 5-17 months
Biological: R78C — A soluble RIPR EGF-CyRPA fusion protein vaccine
  Arms: Group 1(n=8) adults (18-35years); Group 3 (n=8) children aged between 5-17 months; Group 4 (n=8) Children aged between 5-17 months; Group 6 ( n=16) Children 5-17 months
Biological: Matrix-M™ — A saponin-based vaccine adjuvant

SUMMARY:
This is a Phase Ib age de-escalation, dose escalation, open-label study to assess the safety and immunogenicity of the multi-stage malaria vaccine candidate R21 plus RH5.1 and/or R78C in Matrix-M in adults aged 18-35 years and children aged 5-17 months in Burkina Faso.

DETAILED DESCRIPTION:
There will be six study groups. Group 1 will consist of 8 adults who will receive three doses of 5 µg R21 + 10 µg RH5.1 + 10 µg R78C. Group 2 will consist of 8 children who will receive three doses of 5 µg R21 + 10 µg RH5.1. Group 3 will consist of 8 children who will receive three doses of 5 µg R21 + 10 µg R78C. Group 4 will consist of 8 children who will receive three doses of 5 µg R21 + 10 µg RH5.1 +10 µg R78C. Group 5 will consist of 8 children who will receive three doses of 5 µg R21. Group 6 will consist of 16 children who will receive three doses of 10 µg RH5.1 +10 µg R78C. All vaccinations will be given in 50 µg Matrix-M. All groups will receive their vaccinations in a 0-1-6 month regimen.

Groups 1 to 4 and 6 will be recruited in a staggered process. There will be a DSMB review prior to age deescalation. There will also be three sentinel participants per group and DSMB reviews prior to each subsequent (second and third) vaccination. Group 5 can be recruited at any time and without need for sentinel participants or DSMB review.

ELIGIBILITY:
Inclusion Criteria:

Only participants who meet all the inclusion criteria will be enrolled into the trial:

* Group 1: Healthy adult aged 18-35 years at the time of first study vaccination
* Group 2-6: Healthy child aged 5-17 months at the time of first study vaccination
* Group 1: Female participants must be non-pregnant (as demonstrated by a negative urine pregnancy .

test), and practice continuous effective contraception until three months after the final study vaccination

* Participant or parent/guardian provides signed/thumb-printed informed consent
* Participant (and parent/guardian for child participants) resident in the study area villages, and anticipated to be available for vaccination and the duration of follow-up -

Exclusion Criteria:

* The participant may not enter the trial if ANY of the following apply:

  * Clinically significant congenital abnormalities as judged by the PI or other delegated individual.
  * Clinically significant skin disorder (psoriasis, contact dermatitis, etc.), cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness as judged by the PI or other delegated individual.
  * History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
  * Children with weight-for-age Z score of less than -3 or other clinical signs of malnutrition.
  * History of allergic reaction, significant IgE-mediated event, or anaphylaxis to immunisation.
  * History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
  * Sickle cell disease.
  * Clinically significant laboratory abnormality at grade 2 or above as judged by the PI or other delegated individual.
  * Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
  * Receipt of any vaccine in the 14 days preceding enrolment, or planned receipt of any other vaccine within 28 days following each study vaccination.
  * History of vaccination with any malaria vaccine.
  * Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
  * Suspected or known current alcohol misuse.
  * Suspected or known injecting drug use in the 5 years preceding enrolment.
  * Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
  * Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
  * Seropositive for hepatitis B surface antigen (HBsAg), hepatitis C (HCV IgG) or HIV. For children, any history of vertical exposure to HIV infection.
  * Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (for corticosteroids, this will mean prednisone, or equivalent, ≥ 0.5 mg/kg/day; inhaled and topical steroids are allowed).
  * Any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Vaccination and re-vaccination exclusion criteria:

The following adverse events associated with vaccine immunisation constitute absolute contraindications to further administration of vaccine. If any of these events occur during the study, the participant must be withdrawn and followed until resolution of the event, as with any adverse event:

* Anaphylactic reaction following administration of vaccine.
* Pregnancy.

The following adverse events constitute contraindications to administration of vaccine at that point in time; if any one of these adverse events occurs at the time scheduled for vaccination, the participant may be vaccinated at a later date, or withdrawn at the discretion of the Investigator. The participant must be followed until resolution of the event as with any adverse event:

* Acute disease at the time of vaccination (acute disease is defined as the presence of a moderate or severe illness with or without fever or symptoms suggestive of possible COVID-19 disease). All vaccines can be administered to persons with a minor illness such as diarrhoea or mild upper respiratory infection without fever, i.e. axillary temperature < 37.5°C.
* Temperature of >37.5°C (99.5°F) at the time of vaccination.

Ages: 5 Months to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety: To assess the safety and reactogenicity of R21, RH5.1 and R78C in Matrix-M™ when used in different combinations in healthy adults and children living in a malaria-endemic area. | Solicited AEs will be assessed at Day 0, Days 1-6, 28, days 29-34, 182 and days 187. Unsolicited AEs on Day 0, Days 1-6, 14, 28, Days 29-34, 42, 56, 182, Days 183-187 and 196. All SAEs will be assessed throughout the study follow up period upto Day 365
  The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events. The following parameters will be assessed:
  * Occurrence of solicited local reactogenicity signs and symptoms for 7 days following each vaccination (day of vaccination and 6 subsequent days)
  * Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following each vaccination (day of vaccination and 6 subsequent days)
  * Occurrence of unsolicited adverse events for 28 days following the vaccination (day of vaccination and 27 subsequent days)
  * Clinically significant change from baseline for safety laboratory measures throughout the study
  * Occurrence of serious adverse events during the whole study duration.

SECONDARY OUTCOMES:
Immunogenicity: To assess the humoral immunogenicity of R21, RH5.1 and R78C in Matrix-M™ when used in different combinations in healthy adults and children living in a malaria-endemic area. | Immunology blood samples will be collected at screening, day of vaccination, at Days 42, 56, 182, 196, 210, 240, and 365.
  Immunogenicity will be assessed by a variety of immunological assays. The following measures will be assessed:
  * Serum response:
    o Quantitative antigen-specific IgG antibody levels (µg/mL readout) over time - analysis of peak responses and longevity;
  * In vitro GIA against 3D7 clone P. falciparum parasites using purified total IgG and a single-cycle pLDH readout assay

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche en Sciences de la Santé, Siglé, Boulkiemdé Province, Burkina Faso